CLINICAL TRIAL: NCT04461288
Title: Social Media-Based Treatment: Engaging Sexual and Gender Minority Smokers
Brief Title: Engaging Sexual and Gender Minority Cigarette Smokers Into Social Media-based Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Tobacco Related Disease Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRDRP - T29IP0461
Record Dates: First submitted 2020-06-29; First posted 2020-07-08 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Smoking Cessation; Nicotine Dependence; Tobacco Use; Cigarette Smoking
Keywords: smoking; social media; LGBT; sexual and gender minority; nicotine replacement therapy; digital interventions
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder; Tobacco Use; Cigarette Smoking; Smoking; Coitus | interventions — Counseling; Palliative Care; Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Pride Posts (Experimental): This six month intervention will be conducted on the Facebook platform. Participants will receive regular social media posts tailored to the sexual and gender minority communities (LGBTQ+). Weekly live sessions with a tobacco expert will be available. Participants will also have access to up to six months of nicotine replacement therapy (patch + gum/lozenge). Dosage will be based manufacturer's recommendations which are based on self-reported smoking behaviors.
  Interventions: Behavioral: Social media-based education, counseling, and support; Other: Nicotine replacement therapies (NRT)
- Pride Posts Plus (Experimental): This six month intervention will include all elements of the Pride Posts arm. In addition, the intervention will include gamification, gaming elements designed to encourage participation in the program and behavior change. Participants will also have access to up to six months of nicotine replacement therapy (patch + gum/lozenge). Dosage will be based manufacturer's recommendations which are based on self-reported smoking behaviors.
  Interventions: Behavioral: Social media-based education, counseling, and support; Other: Nicotine replacement therapies (NRT); Other: Gamification
- Usual Care Condition (Active Comparator): Participants in this arm will be provided with a referral to smokefree.gov, a federally-funded website which provides support and digital-based interventions to assist in smoking cessation activities. Participants will also have access to up to six months of nicotine replacement therapy (patch + gum/lozenge). Dosage will be based manufacturer's recommendations which are based on self-reported smoking behaviors.
  Interventions: Other: Nicotine replacement therapies (NRT)

INTERVENTIONS:
Behavioral: Social media-based education, counseling, and support — This six-month intervention is culturally-tailored to sexual and gender minority cigarette smokers. The intervention is group-based and includes daily posts and weekly live sessions during the initial three months. Posts and group sessions focus on tobacco use education, developing a quit plan, as well as managing stress, negative thinking, social support, exercise, as techniques to support cessation.
  Arms: Pride Posts; Pride Posts Plus
Other: Nicotine replacement therapies (NRT) — Participants will have access to up to six months of nicotine patch therapy. Participants will start on either 21, 14, or 7 mg patches based on manufacturers recommendations based on smoking behaviors.
  In addition to nicotine patch, participants will have access to a choice of 2 mg. nicotine lozenges or nicotine gum as an adjunct to patch treatment. Participants will be encouraged to use up to 5 pieces daily to address situational urges and cravings for a cigarette.
Other: Gamification — Gaming elements designed to encourage participation in the program and behavior change.
  Arms: Pride Posts Plus

SUMMARY:
This research study will evaluate the preliminary efficacy of Pride Posts Plus, a social media-based smoking cessation treatment. A pilot randomized trial (N=120) will compare Pride Posts Plus, which includes a gamification element, to Pride Posts (without gamification) and to a usual care treatment. Participants will be adults who smoke, identify as sexual or gender minorities, and use Facebook. The primary outcome will be biochemically verified 7-day abstinence from smoking at 3 and 6 months. Secondary outcomes will be treatment engagement, a quit attempt (y/n), and thoughts about tobacco abstinence at 3 and 6 mos.

DETAILED DESCRIPTION:
Participants (N=136) will be randomized to one of three conditions: (1) Pride Posts, a Facebook-delivered smoking cessation intervention (including daily posts, and weekly live group sessions, tailored to sexual and gender minority (SGM) adults; (2) Pride Posts Plus, the Facebook-delivered smoking cessation intervention plus a gamification element, or (2) a usual care condition which includes referral to smokefree.gov, a federally-developed web-based intervention which includes similar digital treatment elements. All participants will have access to up to six months of nicotine replacement therapy (NRT).

Assessments will occur at baseline, 3, and 6 months follow-up. Assessments will include measures on smoking, thoughts about abstinence, and SGM identity experiences. All participants who report no past 7-day smoking will be asked to provide biochemical verification of smoking status using a portable carbon monoxide measurement tool. All intervention and assessment procedures will be conducted digitally.

ELIGIBILITY:
Inclusion Criteria:

* Daily smoker
* Self-identify as sexual and/or gender minority
* Interested in quitting in next 6 months
* 6 months of Facebook experience
* English-speaking

Exclusion Criteria:

* Contraindications to nicotine replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Reported 7-day Biochemically Verified Abstinence at 3 Months | 3 months
  Abstinence is defined by all participants who report no smoking within the last 7 days will use a breathalyzer to measure carbon monoxide levels in the breath to verify smoking abstinence prior to the 3 month assessment.
Number of Participants With Reported 7-day Biochemically Verified Abstinence at 6 Months | 6 months
  Abstinence is defined by all participants who report no smoking within the last 7 days will use a breathalyzer to measure carbon monoxide levels in the breath to verify smoking abstinence prior to the 6 month assessment.

SECONDARY OUTCOMES:
Number of Participants Whom Attempted to Quit Tobacco Use During the Course of Treatment | 3 to 6 months
  Participants will report intentional quit attempts lasting at least 24 hours since treatment initiation or previous assessment
Responses to the Thoughts About Abstinence Questionnaire Over Time | 3 to 6 months
  The Thoughts About Abstinence Questionnaire is a 5 item self-report questionnaire that measures: 1) desire to quit smoking, 2) expected success at quitting, 3) expected difficulty of quitting, and 4) confidence in ability to quit on 10-point Likert scales (e.g., 1=no desire to quit/lowest expectation/lowest level of difficulty to 10 = extreme desire to quit/highest expectation of success/highest expected difficulty.
Frequency of social media posts | 3 to 6 months
  Treatment engagement as measured by frequency of social media posts
Frequency of participation in live group sessions | 3 to 6 months
  Treatment engagement as measured by participation in live group sessions
Duration of Active Participation | 3 to 6 months
  Treatment engagement as measured by duration of active participation in intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Humfleet, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No